CLINICAL TRIAL: NCT05815342
Title: Safety and Efficacy of the Omnipod 5 Automated Insulin Delivery System in Adults With Type 2 Diabetes
Brief Title: OP5-005 Using Omnipod 5 in Adults With Type 2
Acronym: SECURE-T2D
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Insulet Corporation (Industry)
Collaborators: Jaeb Center for Health Research (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: G230013
Record Dates: First submitted 2023-03-21; First posted 2023-04-18 (Actual); Results first posted 2025-09-29 (Actual); Last update posted 2025-09-29 (Actual); Status verified 2025-09

CONDITIONS: Type2 Diabetes
Keywords: T2D; Omnipod; Automated Insulin Delivery

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (1):
- Treatment (Experimental): All subjects wearing the Omnipod 5 Automated Glucose Monitoring System
  Interventions: Device: Omnipod 5 Automated Glucose Control System

INTERVENTIONS:
Device: Omnipod 5 Automated Glucose Control System — The Omnipod Horizon™ Automated Glucose Control System will provide automated insulin delivery

SUMMARY:
This is a single arm, multi-center, prospective study that will evaluate the safety and efficacy of the Omnipod 5 Automated Insulin Delivery System in adults with type 2 diabetes requiring insulin therapy.

DETAILED DESCRIPTION:
This outpatient study consists of 2 phases.

Phase 1 is a 14-day period to collect baseline glucose and insulin data. Participants will manage their diabetes as an outpatient per their usual routine. During this time participants will wear a blinded continuous glucose monitor to collect baseline glycemic information.

Phase 2 is a 13 week treatment period during which participants will use the Omnipod 5 System consisting of the Omnipod 5 pod, Omnipod 5 app as well as a Dexcom G6 continuous glucose monitor. Participants will do in-clinic or virtual visits at least monthly for a total of 8 visits. During the treatment period all participants will undergo supervised exercise and meal challenges.

ELIGIBILITY:
Inclusion Criteria:

1. Age at time of consent 18-75 years
2. Diagnosed with type 2 diabetes, on current insulin regimen for at least 3 months prior to screening (i.e. Basal-bolus, basal only or pre-mix)
3. Basal bolus (long-acting insulin and rapid acting analog) or pre-mix users with A1C <12.0% OR basal users on long or intermediate acting insulin only with A1C > 7.0% and < 12.0%
4. Willing to use only the following types of U-100 insulin during the study: Humalog U-100, Novolog, or Admelog
5. Participant agrees to provide their own insulin for the duration of the study
6. Stable doses over the preceding 4 weeks of other glucose-lowering medications as determined by Investigator
7. Stable doses of weight loss medications over the preceding 4 weeks and throughout the study that may affect glycemic control directly and/or indirectly, except for a dose reduction or discontinuation, as determined by Investigator
8. Willing to wear the system continuously throughout the study
9. Deemed appropriate for pump therapy per investigator's assessment considering previous history of severe hypoglycemic and hyperglycemic events, and other comorbidities
10. Investigator has confidence that the participant has the cognitive ability and can successfully operate all study devices and can adhere to the protocol
11. Able to read and understand English or Spanish
12. Willing and able to sign the Informed Consent Form (ICF)
13. If female of childbearing potential, willing and able to have pregnancy testing

Exclusion Criteria:

1. Use of an AID pump in automated mode within 3 months prior to screening
2. Any medical condition which in the opinion of the investigator, would put the participant at an unacceptable safety risk, such as untreated malignancy, unstable cardiac disease, unstable or end-stage renal disease, and/or eating disorders (i.e. anorexia/bulimia)
3. Current or known history of coronary artery disease that is not stable with medical management, including unstable angina, or angina that prevents moderate exercise despite medical management, or a history of myocardial infarction, percutaneous coronary intervention, or coronary artery bypass grafting within the 12 months prior to screening
4. Any planned surgery during the study which could be considered major in the opinion of the investigator
5. History of more than 1 severe hypoglycemic event in the 6 months prior to screening
6. History of more than 1 episode of diabetic ketoacidosis (DKA) or Hyperosmolar hyperglycemic syndrome (HHS) in the 6 months prior to screening; unrelated to an intercurrent illness; kinked, dislodged, or occluded cannula; or initial diabetes diagnosis
7. Blood disorder or dyscrasia within 3 months prior to screening, including use of hydroxyurea, which in the investigator's opinion could interfere with determination of HbA1c
8. Plans to receive blood transfusion over the course of the study
9. Has taken oral or injectable steroids within 8 weeks prior to screening or plans to take oral or injectable steroids during the study
10. Unable to tolerate adhesive tape or has any unresolved skin condition that could impact sensor or pump placement
11. Pregnant or lactating, planning to become pregnant during the study, or is a woman of childbearing potential and not on acceptable form of birth control (acceptable includes abstinence, condoms, oral/injectable contraceptives, IUD, or implant); childbearing potential means that menstruation has started, and the participant is not surgically sterile or greater than 12 months post-menopausal)
12. Participation in another clinical study using an investigational drug or device other than the Omnipod 5 in the 30 days prior to screening or intends to participate during the study period
13. Unable to follow clinical protocol for the duration of the study or is otherwise deemed unacceptable to participate in the study per the investigator's clinical judgment
14. Participant is an employee of Insulet, an Investigator or Investigator's study team, or immediate family member (spouse, biological or legal guardian, child, sibling, parent) of any of the aforementioned

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 343 (Actual)
Dates: Start 2023-04-11 (Actual); Primary Completion 2024-03-01 (Actual); Study Completion 2024-03-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Francisco J Pasquel, MD, Study Chair — Emory School of Medicine
Locations (21):
- United States (21):
  - University of Southern California, Los Angeles, California
  - Sansum Diabetes Research Institute, Santa Barbara, California
  - University of Colorado, Aurora, Colorado
  - East Coast Institute for Research, Jacksonville, Florida
  - Metabolic Research Institute, West Palm Beach, Florida
  - Emory, Atlanta, Georgia
  - East Coast Institute for Research, Canton, Georgia
  - Endocrine Research, Roswell, Georgia
  - Joslin Diabetes, Boston, Massachusetts
  - Henry Ford, Detroit, Michigan
  - Health Partners, Minneapolis, Minnesota
  - Albert Einstein College of Medicine, The Bronx, New York
  - MAHEC, Asheville, North Carolina
  - University of North Carolina, Chapel Hill, North Carolina
  - Physicians East, Greenville, North Carolina
  - AccellaCare, Wilmington, North Carolina
  - Ohio State, Columbus, Ohio
  - University Diabetes and Endocrine Consultants, Chattanooga, Tennessee
  - Texas Diabetes and Endocrinology, Austin, Texas
  - Diabetes and Thyroid Center, Fort Worth, Texas
  - Diabetes and Glandular Disease Clinic, San Antonio, Texas

REFERENCES:
- [Derived] Pasquel FJ, Davis GM, Huffman DM, Peters AL, Parker JC, Laffel LM, Romeo GR, Mathew J, Castorino KN, Kruger DF, Dungan KM, Kipnes M, Jauch EC, Oser TK, Shah VN, Horowitz B, Carlson AL, Warren ML, Deeb W, Buse JB, Reed JH, Berner J, Blevins T, Bajaj C, Kollman C, Raghinaru D, Ly TT, Beck RW; Omnipod 5 SECURE-T2D Consortium. Automated Insulin Delivery in Adults With Type 2 Diabetes: A Nonrandomized Clinical Trial. JAMA Netw Open. 2025 Feb 3;8(2):e2459348. doi: 10.1001/jamanetworkopen.2024.59348. PMID 39951268

RESULTS

PARTICIPANT FLOW:
Period: Baseline, Standard Therapy (2 Weeks)
Arm/Group | Treatment
Started | 320
Completed | 305
Not Completed | 15
Not completed — Ineligible | 4
Not completed — Withdrawal by Subject | 9
Not completed — Lost to Follow-up | 2
Period: Treatment Phase (13 Weeks)
Arm/Group | Treatment
Started | 305
Completed | 289
Not Completed | 16
Not completed — Withdrawal by Subject | 14
Not completed — Lost to Follow-up | 2

BASELINE CHARACTERISTICS:
Arm/Group | Treatment
Number analyzed (Participants) | 305
Age, Continuous [Mean (Standard Deviation); unit: years] | 57 (11)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 175
  Male | 130
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  American Indian or Alaskan Native, not Hispanic or Latino | 2
  Asian or Pacific Islander, not Hispanic or Latino | 7
  Black, not Hispanic or Latino | 72
  Hispanic or Latino | 66
  White, not Hispanic or Latino | 153
  ≥1 Race, not Hispanic or Latino | 3
  Unknown | 2
BMI [Mean (Standard Deviation); unit: kg/m^2] | 35 (8)
HbA1C [Mean (Standard Deviation); unit: Percentage of HbA1C] | 8.2 (1.3)

OUTCOME MEASURES:

1. Primary Outcome: Change in HbA1c
Description: The change in HbA1c at 13 weeks from baseline
Time Frame: Comparing the change in HbA1c during the 13 weeks study phase
Population: The number of participants with available data ranged from 294 to 305 across outcomes.
Measure: Mean (Standard Deviation); unit: Percentage of HbA1C
Arm/Group | Treatment
Number analyzed (Participants) | 296
Percentage of HbA1C
  Baseline or Standard Therapy (2 weeks) | 8.2 (1.3)
  End of treatment or treatment phase (13 weeks) | 7.4 (0.9)

2. Secondary Outcome: Mean Glucose
Description: Glucose metric from study provided continuous glucose monitor (CGM)
Time Frame: Measuring mean glucose during the 13 weeks study phase
Population: Based on the pre-specified criteria ("CGM analyses will include all participants with ≥168 hours of CGM data during each of the Standard therapy period and the 13-week treatment period."), N=299 for the glycemic metrics.
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Treatment
Number analyzed (Participants) | 299
mg/dL
  Baseline or Standard Therapy (2 weeks) | 202 (50)
  End of treatment or treatment phase (13 weeks) | 170 (24)

3. Secondary Outcome: Percentage of Time in Range 70-180 mg/dL
Description: Glucose metric from CGM
Time Frame: Measured during 13 weeks study phase
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Percent Time in Range
Arm/Group | Treatment
Number analyzed (Participants) | 299
Percent Time in Range
  Baseline or Standard Therapy (2 weeks) | 45 (25)
  End of treatment or treatment phase (13 weeks) | 66 (17)

4. Secondary Outcome: Percent of Time in Range 70-140 mg/dL
Description: Glucose metric from study CGM
Time Frame: Measured during 13 weeks study phase
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Percent Time in Range
Arm/Group | Treatment
Number analyzed (Participants) | 299
Percent Time in Range
  Baseline or Standard Therapy (2 weeks) | 21 (18)
  End of treatment or treatment phase (13 weeks) | 33 (17)

5. Secondary Outcome: Percent of Time ≥ 300 mg/dL
Description: Glucose metric from CGM
Time Frame: Measured during 13 weeks study phase
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Percent Time in Range
Arm/Group | Treatment
Number analyzed (Participants) | 299
Percent Time in Range
  Baseline or Standard Therapy (2 weeks) | 7.9 (10.3)
  End of treatment of treatment phase (13 weeks) | 7.9 (2.4)

6. Secondary Outcome: Percent of Time > 250 mg/dL
Description: Glucose metric from CGM
Time Frame: Measured during 13 weeks study phase
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Percent Time in Range
Arm/Group | Treatment
Number analyzed (Participants) | 299
Percent Time in Range
  Baseline or Standard Therapy (2 weeks) | 20 (22)
  End of treatment or treatment phase (13 weeks) | 7 (8)

7. Secondary Outcome: Percent of Time >180 mg/dL
Description: Glucose metric from CGM
Time Frame: Measured during 13 weeks study phase
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Percent Time in Range
Arm/Group | Treatment
Number analyzed (Participants) | 299
Percent Time in Range
  Baseline or Standard Therapy (2 weeks) | 54 (25)
  End of treatment or treatment phase (13 weeks) | 34 (17)

8. Secondary Outcome: Percent of Time < 70 mg/dL [Non-inferiority; Non-inferiority Limit 2.0%]
Description: Glucose metric from CGM
Time Frame: Measured during 13 weeks study phase
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Percent Time in Range
Arm/Group | Treatment
Number analyzed (Participants) | 299
Percent Time in Range
  Baseline or Standard Therapy (2 weeks) | 0.2 (0.3)
  End of treatment or treatment phase (13 weeks) | 0.2 (0.2)

9. Secondary Outcome: Percent of Time < 54 mg/dL [Non-inferiority; Non-inferiority Limit 0.5%]
Description: Glucose metric from CGM
Time Frame: Measured during 13 weeks study phase
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Percent Time in Range
Arm/Group | Treatment
Number analyzed (Participants) | 299
Percent Time in Range
  Baseline or Standard Therapy (2 weeks) | 0.01 (0.02)
  End of treatment or treatment phase (13 weeks) | 0.04 (0.05)

10. Secondary Outcome: Change From Baseline in T2-DDAS Total Score
Description: A questionnaire that measures seven critical dimensions of distress (28-item scale with 6 choices that range from 1 (Not a Problem) to 6 (A Very Serious Problem)). The total score can range from 1 to 6, with a lower score indicating a better outcome.
Time Frame: Baseline compared to end of week 13 visit
Measure: Mean (Standard Deviation); unit: Score
Arm/Group | Treatment
Number analyzed (Participants) | 305
Score
  Baseline or Standard Therapy (2 weeks) | 2.5 (1.0)
  End of treatment or treatment phase (13 weeks) | 2.2 (0.9)

11. Secondary Outcome: Percentage Meeting MCID for T2-DDAS
Description: as for outcome 10
Time Frame: Baseline compared to end week 13 visit
Measure: Number; unit: Percentage
Arm/Group | Treatment
Number analyzed (Participants) | 299
Percentage
  Baseline or Standard Therapy (2 weeks) | 66
  End of treatment or treatment phase (13 weeks) | 55

12. Secondary Outcome: Change From Baseline in Pittsburgh Sleep Quality Index Total Score
Description: Change from baseline in PSQI total score which assesses sleep quality over a one month interval. The survey includes 10 self-rated items.
  Minimum Score = 0 (better); Maximum Score = 21 (worse). Lower scores indicate better outcomes (eg, less distress related to diabetes, better sleep quality).
Time Frame: Baseline compared to end of week 13 visit
Population: The number of participants with available data ranged from 294 to 305 across outcomes.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Treatment
Number analyzed (Participants) | 305
score on a scale
  Baseline or ST (2 weeks): number analyzed (Participants) | 304
  Baseline or ST (2 weeks) | 7.3 (4.0)
  End of treatment or treatment phase (13 weeks): number analyzed (Participants) | 294
  End of treatment or treatment phase (13 weeks) | 7.0 (4.1)

13. Secondary Outcome: % Meeting MCID for Pittsburgh Sleep Quality Index
Description: Change from baseline in PSQI total score which assesses sleep quality over a one month interval. The survey includes 10 self-rated items.
Time Frame: Baseline compared to end of week 13 visit
Population: The number of participants with available data ranged from 294 to 305 across outcomes.
Measure: Number; unit: Percentage
Arm/Group | Treatment
Number analyzed (Participants) | 305
Percentage
  Baseline or ST (2 weeks): number analyzed (Participants) | 304
  Baseline or ST (2 weeks) | 63
  End of treatment or treatment phase (13 weeks): number analyzed (Participants) | 294
  End of treatment or treatment phase (13 weeks) | 59

14. Secondary Outcome: Change From Baseline in HCS Total Score
Description: Questionnaire that examines the degree to which people with diabetes feel able, secure, and comfortable regarding their ability to stay safe from hypoglycemic-related problems (9-item scale with 4 choices that range from 1 (Not Confident At All) to 4 (Very Confident)). The total score can range from 1 to 4, with a higher score indicating a better outcome.
Time Frame: Baseline compared to end week 13 visit
Population: The number of participants with available data ranged from 294 to 305 across outcomes.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Treatment
Number analyzed (Participants) | 305
score on a scale
  Baseline of Standard Therapy (2 weeks) | 3.2 (0.6)
  End of treatment or treatment phase (13 weeks): number analyzed (Participants) | 300
  End of treatment or treatment phase (13 weeks) | 3.3 (0.6)

15. Secondary Outcome: % Meeting MCID for HCS
Description: as for outcome 14
Time Frame: Baseline compared to end week 13 visit
Population: The number of participants with available data ranged from 294 to 305 across outcomes.
Measure: Number; unit: Percentage
Arm/Group | Treatment
Number analyzed (Participants) | 305
Percentage
  Baseline or Standard Therpey (2 weeks) | 32
  End of treatment or treatment phase (13 weeks): number analyzed (Participants) | 300
  End of treatment or treatment phase (13 weeks) | 0.2

16. Secondary Outcome: Percentage of Time <70 mg/dL (Superiority)
Description: Glucose metric from CGM
Time Frame: Measured during 13 weeks study phase
Population: The number of participants with available data ranged from 294 to 305 across outcomes.
Measure: Mean (Standard Deviation); unit: Percent Time in Range
Arm/Group | Treatment
Number analyzed (Participants) | 305
Percent Time in Range
  Baseline or Standard Therapy (2 weeks) | 0.2 (0.3)
  End of treatment or treatment phase (13 weeks) | 0.2 (0.2)

17. Secondary Outcome: Percentage of Time <54 mg/dL (Superiority)
Description: Glucose metric from CGM
Time Frame: Measured during 13 weeks study phase
Population: The number of participants with available data ranged from 294 to 305 across outcomes.
Measure: Mean (Standard Deviation); unit: Percent Time in Range
Arm/Group | Treatment
Number analyzed (Participants) | 305
Percent Time in Range
  Baseline or ST (2 weeks) | 0.01 (0.02)
  End of treatment or treatment phase (13 weeks) | 0.04 (0.05)

18. Secondary Outcome: Coefficient of Variation
Description: Glucose metric from study continuous glucose monitoring system (CGM)-measured glucose variability with the coefficient of variation (CV). Calculated by dividing the standard deviation of CGM values by the mean CGM values in the observation period.
Time Frame: Measured during 13 weeks study phase and compared to standard therapy
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Percent coefficient of variation
Arm/Group | Treatment
Number analyzed (Participants) | 299
Percent coefficient of variation
  Baseline or Standard Therapy (2 weeks) | 27.8 (6.3)
  End of treatment or treatment phase (13 weeks) | 27.1 (5.1)

ADVERSE EVENTS:
Time Frame: Adverse events were collected from the start of standard therapy until the end of the 13-week treatment phase.
Groups:
- Standard Therapy: Adverse events collected during the 2-week Baseline or Standard Therapy Phase.
- Treatment: Adverse events collected during the 13-week treatment phase while wearing the Omnipod 5 Automated Glucose Monitoring System
  Omnipod 5 Automated Glucose Control System: The Omnipod Horizon™ Automated Glucose Control System will provide automated insulin delivery
Arm/Group | Standard Therapy | Treatment
All-Cause Mortality (participants affected / at risk) | 0/320 | 0/305
Serious Adverse Events (participants affected / at risk) | 1/320 | 13/305
Other Adverse Events (participants affected / at risk) | 3/320 | 43/305
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Standard Therapy (N=320) | Treatment (N=305)
Severe hypoglycemia (Endocrine disorders) | 1 (1) | 0 (0)
Nonglycemic serious adverse events (General disorders) | 0 (0) | 13 (13)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Standard Therapy (N=320) | Treatment (N=305)
Nonserious adverse event (Gastrointestinal disorders) | 3 (3) | 43 (53)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2024-02-27): https://cdn.clinicaltrials.gov/large-docs/42/NCT05815342/Prot_SAP_000.pdf